CLINICAL TRIAL: NCT00214552
Title: A Double-blind Placebo Controlled Clinical Trial to Evaluate the Effects on Asthma Control of Rabeprazole Given Twice Daily in Subjects With Asthma.
Brief Title: Evaluate the Effects on Asthma Control of Rabeprazole Given Twice Daily in Subjects With Asthma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Associated Scientists to Help Minimize Allergies (Other)
Collaborators: Janssen Pharmaceuticals (Industry); Eisai Inc. (Industry)
Responsible Party: Stephen A Tilles, MD, Principal Investigator, ASTHMA, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RAB-USA-38
Record Dates: First submitted 2005-09-10; First posted 2005-09-22 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Asthma; Gastroesophageal Reflux Disease
Keywords: GERD; Gastroesophageal reflux disease; Asthma symptoms
MeSH Terms: conditions — Asthma; Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rabeprazole

SUMMARY:
The hypothesis for this study is that potent anti-secretory therapy with high dose PPI improves asthma control regardless of either asthma severity or the presence of GERD symptoms.

DETAILED DESCRIPTION:
Many patients with GERD do not experience heartburn symptoms. Barium esophagram, endoscopy and/or overnight esophageal pH monitoring are commonly relied upon to objectively establish the diagnosis of GERD. In general, overnight esophageal pH monitoring is the most sensitive and specific test available to confirm GERD. However, the literature exploring GERD as a cause of chronic cough suggests that the currently accepted criteria for defining abnormal overnight esophageal pH may not be adequately sensitive. It is therefore possible that aggressive GERD therapy may improve asthma control in patients with "normal" overnight esophageal pH probe results. To our knowledge, there are no published data addressing this question.

Primary Objective The primary objective is to compare asthma control in asthmatic subjects treated with high dose PPI with asthmatic subjects taking placebo PPI. The primary outcome variables will be measurements of asthma symptoms and asthma quality of life.

Secondary Objectives Secondary objectives include evaluating the effect of this aggressive anti-secretory therapy on lung function, asthma medication use (including both baseline and rescue medication), and GERD symptoms. An additional secondary objective will be to evaluate whether the presence or absence of GERD symptoms at baseline (prior to proton pump inhibitor therapy) will independently associate with improvement in any of the other outcomes measured.

Measurements will include: Juniper Asthma Control Questionnaire (visits 2 and 5), Juniper Asthma Quality of Life Questionnaire (visits 2 - 5), GSAS gastroesophageal reflux instrument (visit 2, visit 5), the occurrence of adverse events, change in FVC, FEF25-75%, MIF50 / MEF50, peak expiratory flow rate, FEV1 reversibility, and the physical exam.

Additional measurements will include methacholine challenge and eosinophilia in induced sputum specimens. Induced sputum will be offered to all patients, though it is anticipated that only approximately 50% will agree to this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be 18 years of age or older.
* Subjects baseline FEV1 must be greater than or equal to 50% of predicted at both Visit 1 and visit 2, when all bronchodilators medications have been withheld for the specified intervals.
* Subjects must have physician-diagnosed asthma at visit 1 and report ongoing chronic or intermittent symptoms that include at least one of the following: wheezing, chest tightness, dyspnea, or cough.
* All subjects with a baseline FEV1 greater than or equal to 70% predicted must have a positive methacholine challenge (provocative dose required to reduce FEV1 20% is less than or equal to 10 mg inhaled methacholine) at either visit 1 or visit 2.
* All subjects with a baseline FEV1 greater than 50% but less than 70% must demonstrate at least 12% improvement in FEV1 after a bronchodilator is administered at visit 1 or visit 2.
* Subjects must report using rescue inhaled beta adrenergic agonist treatment at least twice weekly for asthma symptoms (e.g. 2 or more nebulized treatments or 4 or more puffs of inhaled albuterol per week).
* Subjects must experience asthma symptoms (wheezing, shortness of breath, cough, chest tightness, or nocturnal awakening) of at least mild severity on at least 2 days out of each week of run-in (1 week equals 7 days). In addition, the asthma symptom diary card score (over a two week period) must total at least 10 as recorded by the study subject in the run-in diary card. The run-in period may vary in length from 7 days to 28 days, as long as the 10 point score is achieved in a 10 day period.
* Subjects must be free of any clinically significant disease other than asthma.
* Women of childbearing potential must have a negative urine (hCG) pregnancy test at visit 1 or visit 2 and agree, if sexually active, to use medically accepted contraception as defined in ICH guidelines throughout the study.
* Subjects must agree to have the investigator inform their usual treating physician (if other than the study investigator) of their participation in the study.

Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* Subjects who have required daily or alternate day oral corticosteroid treatment for more than a total of 21 days during the 6 months immediately prior to Visit 1.
* Subjects who require daily treatment with proton pump inhibitors, H2-receptor antagonists, or OTC anti-reflux medications).
* Subjects on immunotherapy, unless they are on a stable maintenance schedule for at least 6 months.
* Subjects who have used any investigational drug in the 30 days prior to visit 1.
* Subjects who have experienced allergic or idiosyncratic reactions to PPI, corticosteroid, or inhaled beta adrenergic agonist agents.
* Subjects demonstrating a change in FEV1 of 20% or more between visit 1 and 2.
* Subjects who have required ventilatory support for respiratory failure due to asthma within 5 years of Visit 1.
* Subjects who smoke, have smoked within the past 6 months, or have more than a 15 pack-year history of smoking.
* Subjects who have required hospitalization for asthma in the previous 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2002-09; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Asthma symptoms

SECONDARY OUTCOMES:
Asthma quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Tilles,, MD, Principal Investigator — ASTHMA, Inc.
Locations (2):
- United States (2):
  - ASTHMA, Inc., Richland, Washington
  - ASTHMA, Inc., Seattle, Washington